CLINICAL TRIAL: NCT00234000
Title: A Phase I Multicenter Study of Arsenic Trioxide and Azacitidine in Patients With Myelodysplastic Syndromes
Brief Title: Azacitidine and Arsenic Trioxide in Treating Patients With Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was closed due to poor enrollment
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: CTI BioPharma (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000442931; UCLA-0408087
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2012-08

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; refractory anemia with ringed sideroblasts; refractory anemia; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory; Leukemia, Myelomonocytic, Chronic | interventions — Arsenic Trioxide; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): see description in intervention
  Interventions: Drug: arsenic trioxide; Drug: azacitidine

INTERVENTIONS:
Drug: arsenic trioxide — Each 28-day treatment cycle will include dosing for 2 days per week of ATO. Subjects will recieve 1 mg/mL each dosing day.
  Other Names: ATO
Drug: azacitidine — Each 28-day treatment cycle will include dosing the first five days of cycle with Azacitidine. Cohorts of three to six patients will each receive 25, 50, and 75 mg/m2/d injected subcutaneously.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as azacitidine and arsenic trioxide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of azacitidine when given together with arsenic trioxide and to see how well they work in treating patients with myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of azacitidine when given in combination with arsenic trioxide in patients with myelodysplastic syndromes (MDS). (Phase I)
* Determine the safety and tolerability of this regimen in these patients. (Phase I)
* Determine the major hematologic response (erythroid response) rate in patients with transfusion-dependent lower-risk MDS treated with this regimen. (Phase II)
* Determine complete and partial remission rates in patients with higher-risk MDS treated with this regimen. (Phase II)
* Determine the toxicity profile of this regimen in these patients. (Phase I)

Secondary

* Determine time to disease progression in patients treated with this regimen. (Phase I and II)
* Determine the overall and progression-free survival of patients treated with this regimen. (Phase I and II)

OUTLINE: This is an multicenter, open-label, phase I, dose escalation study of azacitidine followed by a phase II study. Patients enrolled in the phase II portion are stratified according to baseline International Scoring System score (lower-risk myelodysplastic syndromes [MDS] vs higher-risk MDS).

* Phase I: Patients receive azacitidine subcutaneously once daily on days 1-5 and arsenic trioxide IV over 1-4 hours on days 1, 4, 8, 11, 15, 18, 22, and 25. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with stable disease may receive up to 8 courses of therapy. Patients with responding disease may continue to receive study therapy until a major response or a complete remission is achieved.

Cohorts of 3-6 patients receive escalating doses of azacitidine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive arsenic trioxide as in phase I and azacitidine as in phase I at one dose level below the MTD determined in phase I.

After the completion of study treatment, patients are followed at 4 weeks and then every 3-12 months for survival.

PROJECTED ACCRUAL: Approximately 3-18 patients will be accrued for the phase I portion of this study. A total of 60 patients (30 per stratum) will be accrued for the phase II portion of this study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MDS by standard criteria. Patients within each of the FAB diagnostic groups of RA, RARS, RAEB, RAEBt, and CMML are eligible. For patients with lower-risk MDS only: documented red blood cell dependence, defined as the inability to maintain a hematocrit of > 25% without transfusion support.
* Adequate marrow iron stores
* In patients with serum erythropoietin less than 200 IU/mL at screening, failure to have responded to a 2 to 3 month trial of recombinant erythropoietin
* Serum creatinine or serum bilirubin < 1.5 times the upper limit of normal; higher levels are acceptable if ALT levels < 2 x upper limits of normal
* Women of childbearing potential must have a negative serum pregnancy test prior to azacitidine/treatment.
* Women of childbearing potential should be advised to avoid becoming pregnant and should be advised to not father a child while receiving treatment with azacitidine
* Age > 18 years

Exclusion Criteria:

* Treatment with growth factors within the 30 days before first treatment with ATO/Azacitidine, except that patients with serum erythropoietin < 200 IU/mL who failed to respond to a trial with EPO are not excluded regardless of the time since last EPO
* Treatment with cytotoxic or experimental agents within 30 days before first treatment with ATO/Azacitidine
* Absolute QT interval > 460 msec in the presence of adequate serum potassium and magnesium values
* Active serious infections that are not controlled by antibiotics
* Pregnant or lactating women
* Inability or unwillingness to comply with the treatment protocol, follow-up, or research tests
* NYHA Class III or IV heart failure
* Poorly controlled hypertension, diabetes mellitus, or other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-02; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by NCI CTCAE v3.0 (Phase I) | Every 28 days upto 8 months

SECONDARY OUTCOMES:
Time to disease progression | Participants are folowed for an average of 1 year after completion of study treatment
Overall survival | Participants are followed every 3-12 months for survival

CONTACTS AND LOCATIONS:
Overall Officials: Gary J. Schiller, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States